CLINICAL TRIAL: NCT01028443
Title: Efficacy of Topical Cyclosporine A for Treatment and Prevention of Graft Rejection in Corneal Grafts With Previous Rejection Episodes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8546
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2006-04

CONDITIONS: Endothelial Graft Rejection
MeSH Terms: interventions — Cyclosporine

ARMS (2):
- Cyclosporine A 2% (Active Comparator)
  Interventions: Drug: Sandimmune
- Artificial tears (Placebo Comparator)
  Interventions: Drug: Artelose

INTERVENTIONS:
Drug: Sandimmune
  Arms: Cyclosporine A 2%
Drug: Artelose
  Arms: Artificial tears

SUMMARY:
The use of topical Cyclosporine A early after an episode of endothelial graft rejection after penetrating keratoplasty and continuing its administration for 6 months can reduce the course of that episode and recurrence of the rejection.

ELIGIBILITY:
Inclusion Criteria:

* Penetrating keratoplasty in eyes without vascularization

Exclusion Criteria:

* History of previous intraocular surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The rate of rejection after drop sessation | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran